CLINICAL TRIAL: NCT06450548
Title: Dynamic 68Ga-PSMA and 18F-FDG PET/CT Analysis of Metastatic Prostatic Adenocarcinomas Prior to 177Lu-PSMA Treatment
Brief Title: Dynamic 68Ga-PSMA and 18F-FDG PET/CT Analysis Prior to 177Lu-PSMA
Acronym: PYPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB23.04
Record Dates: First submitted 2024-05-28; First posted 2024-06-10 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer Metastatic
Keywords: prostate cancer; 68GA-PSMA; parametric acquisition
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic and static acquisition (Experimental): Dynamic and static PET acquisitions with 18F-FDG and 68Ga-PSMA will be performed with a minimum of 24 hours and a maximum of 15 days between the two
  Interventions: Other: Parametric acquisition

INTERVENTIONS:
Other: Parametric acquisition — Parametric acquisition for 18F-FDG PET/CT and 68GA-PSMA PET/CT with 24 h at 15 days of interval

SUMMARY:
Prostate cancer is a significant health issue, representing 21.8% of male cancer cases in France with over 449,000 new cases in 2018. It's the cause of 10% of cancer deaths in Europe.

The PSMA is a target for mCRPC treatment, with therapies like 177Lu-PSMA-617 delivering radiation to cancer cells. The Vision study showed that 177Lu-PSMA-617, combined with standard care, improved survival rates significantly compared to standard care alone.The French ANSM authorized 177Lu-PSMA-617 for mCRPC under certain conditions. Patients must have histologically confirmed mCRPC, be progressive despite treatment, and have PSMA-positive imaging.

Imaging assessments include PSMA PET/CT and 18F-FDG PET/CT to identify FDG-positive and PSMA-negative sites, which are associated with a poorer prognosis.

Parametric analysis using dynamic PET could improve lesion characterization, aiding in treatment decisions. This is the focus of the PyPET study.

The main objective focuses on a comparative analysis of data from dynamic parametric analysis (metabolic influx rate Ki, volume of distribution Vd) and static analysis (standard at 1 hour) using 18F-FDG and 68Ga-PSMA PET/CT for diagnosing metastases, especially in the liver, lymph nodes, and bones. It aims to assess the effectiveness of these imaging techniques in accurately identifying metastatic sites.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Progressive metastatic castration-resistant prostate adenocarcinoma, which has been treated with taxane chemotherapy and at least one anti-androgen hormone therapy.
* Evaluated by 18F-FDG and 68Ga-PSMA PET/CT prior to potential treatment with 177Lu-PSMA.
* Affiliated with or beneficiary of a social protection scheme.
* WHO stage 0 or 1.

Exclusion Criteria:

* Patients unable to understand the study for any reason or comply with the trial requirements (due to language barriers, psychological issues, geographical constraints, etc.).
* Patients unable to undergo the examinations and/or maintain a prolonged lying position (due to back pain, etc.).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2028-03-05 (Estimated); Study Completion 2028-03-05 (Estimated)

PRIMARY OUTCOMES:
Comparative analysis of data from dynamic parametric analysis (volume of distribution Vd) and static analysis | 15 days
Comparative analysis of data from dynamic parametric analysis (metabolic influx rate Ki) and static analysis | 15 days

SECONDARY OUTCOMES:
compare the number of lesions detected as PSMA positive/negative and FDG positive/negative | 15 days
  Comparison of the number of lesions detected as PSMA positive/negative and FDG positive/negative through factorial analysis versus the visual analysis obtained from dynamic and static images (results from the main objective analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Decazes, MD,PhD, Study Director — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France